CLINICAL TRIAL: NCT01433666
Title: Effects of Roflumilast on Cognition in Healthy Adults: a Behaviour-EEG Study
Brief Title: Roflumilast and Cognition
Acronym: EEGrofl
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: METC11-3-035; ZonMw (the Netherlands) (Other Grant/Funding Number: 95110091); 2011-002070-23 (EudraCT Number)
Record Dates: First submitted 2011-06-27; First posted 2011-09-14 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2013-09

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Roflumilast; Phosphodiesterase 4 Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- roflumilast 100ug (Experimental)
  Interventions: Drug: roflumilast (EU: Daxas, USA: Daliresp); Drug: roflumilast
- roflumilast 300ug (Experimental)
  Interventions: Drug: roflumilast (EU: Daxas, USA: Daliresp); Drug: roflumilast
- roflumilast1000ug (Experimental)
  Interventions: Drug: roflumilast (EU: Daxas, USA: Daliresp); Drug: roflumilast
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: roflumilast

INTERVENTIONS:
Drug: roflumilast (EU: Daxas, USA: Daliresp) — Acute intervention: 1 time each dose on different days. Capsulated
  Arms: roflumilast 100ug; roflumilast 300ug; roflumilast1000ug
Drug: Placebo — Acute intervention: single administration, capsulated form.
  Arms: placebo
Drug: roflumilast — Acute intervention: 1 time each dose (100ug, 300ug, 1000ug, placebo). Capsulated.
  Other Names: Daxas; Daliresp; PDE4-inhibitor

SUMMARY:
The aim of the current project is to validate PDE4 inhibitors as a target for cognition enhancers (proof-of-concept) using a translational behaviour-EEG approach. The project will demonstrate whether memory, but also attention, information processing or executive function improves with the PDE4 inhibitor roflumilast in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 years of age
* Healthy (i.e. absence of all exclusion criteria), normal static binocular acuity (corrected or uncorrected),
* Body mass index between 18.5 and 30
* Willingness to sign an informed consent.
* Positive evaluation on the memory screening

Exclusion Criteria:

* History of cardiac, hepatic, renal, pulmonary, neurological, gastrointestinal, haematological, or psychiatric illness
* First-degree relative with psychiatric disorder (in particular major depressive disorder and suicidality)
* Excessive drinking (>20 glasses of alcohol containing beverages per week)
* Pregnancy or lactation
* Use of chronic medication other than oral contraceptives
* Use of recreational drugs in the 2 weeks preceding participation
* Smoking
* Orthostatic hypotension
* Lactose intolerance
* Sensory or motor deficits which could reasonably be expected to affect test performance

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of words remembered on Verbal learning task | 1hr after drug intake
  30 monosyllable words will be displayed on a computer screen. Immediately after the presentation and after 45 minutes, subjects will be asked to report as much words as they remember. In addition, a recognition trial is conducted. Here, 30 words will be presented; 15 new words and 15 from the original list. Subjects have to indicate whether the word is old or new.

CONTACTS AND LOCATIONS:
Overall Officials: Jos H. Prickaerts, PhD, Study Director — Maastricht University
Locations (1):
- Maastricht University, Faculty of Psychology and Neuroscience, Maastricht, Limburg, Netherlands

REFERENCES:
- [Result] Heckman PRA, Van Duinen MA, Blokland A, Uz T, Prickaerts J, Sambeth A. Acute administration of roflumilast enhances sensory gating in healthy young humans in a randomized trial. Psychopharmacology (Berl). 2018 Jan;235(1):301-308. doi: 10.1007/s00213-017-4770-y. Epub 2017 Nov 3. PMID 29098341
- [Result] Van Duinen MA, Sambeth A, Heckman PRA, Smit S, Tsai M, Lahu G, Uz T, Blokland A, Prickaerts J. Acute administration of roflumilast enhances immediate recall of verbal word memory in healthy young adults. Neuropharmacology. 2018 Mar 15;131:31-38. doi: 10.1016/j.neuropharm.2017.12.019. Epub 2017 Dec 11. PMID 29241652
- See also: Published sensory gating data — https://link.springer.com/article/10.1007%2Fs00213-017-4770-y